CLINICAL TRIAL: NCT05099562
Title: Precision Acupuncture in the Treatment of Peripheral Neuropathy After Taxanes Chemotherapy in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHQU-2021005
Record Dates: First submitted 2021-09-27; First posted 2021-10-29 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: acupuncture; breast cancer; peripheral neuropathy; taxane chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture group (Experimental): This is a one-arm study. Breast cancer patients with peripheral neuropathy were measured using the FACT/ GOG-Ntx and EORTC QLQ-CIPN20 scales. Our clinical study included breast cancer patients diagnosed with peripheral neurotoxicity caused by taxanes-based drugs who would receive acupuncture treatment. Neurotoxicity was identified based on NCI-CTCAE 5.0 for daily or almost daily numbness in the hands and feet, tingling, and other symptoms of peripheral neuropathy over the past two to three weeks. Blood samples were collected from patients to detect SNP associated with neurotoxicity.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Patients received standardized acupuncture treatment. A blood sample of genomic DNA storage was taken from the back of the hand between the first and second metacarpals. Genotypes were obtained by oligonucleotide ligation/polymerase chain reaction and capillary electrophoresis of peripheral neuropathy-associated SNPs.

SUMMARY:
Precision Acupuncture in the Treatment of Peripheral Neuropathy After Taxane Chemotherapy in Breast Cancer

DETAILED DESCRIPTION:
Associated peripheral neuropathy in breast cancer patients has a significant impact on their quality of life and treatment compliance. Many studies have shown that acupuncture has a certain therapeutic effect on peripheral neuropathy. Studies have shown that taxane induced peripheral neuropathy in breast cancer is related to genetic factors. Based on SNPs related to peripheral neuropathy, this study screened SNPs related to peripheral neuropathy caused by taxane drugs, and established a prognostic model.

Eligible patients diagnosed with stage I, II or IIIA breast cancer and experiencing peripheral neuropathy for at least 2 weeks were assessed by the Functional Assessment of Cancer Therapy/Gynaecologic Oncology Group-Neurotoxicity，FACT/GOG-Ntx) and the European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire-CIPN twenty-item scale(EORTC QLQ-CIPN20). Likert level 5 and level 4 scores were used for all items in the above two scales. The investigators will temporarily divide the study into a group, and the investigators will increase the group if necessary. Laboratory personnel were blinded to all clinical and outcome data.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was at least 18 years old and had reported grade 1 or higher neuropathic symptoms for more than 2 weeks;
2. Patients were screened for eligibility by the investigator prior to enrollment, including verification of baseline neuropathic symptoms.
3. Patients had a diagnosis of stage I, II, or IIIA breast cancer;
4. Have completed at least 2 weeks of chemotherapy;
5. Higher scores indicate more severe symptoms;
6. Voluntarily participate in the clinical trial and sign the informed consent form after informed consent (patients voluntarily accept the treatment and give informed consent);
7. Eastern Cooperative Oncology Group (ECOG ) score of physical condition (0-1);
8. Patients with previous local recurrence were eligible;
9. The basic indexes were consistent, and the blood routine and ECG were normal.

Exclusion Criteria:

1. patients with needle phobia;
2. Low platelet count (<50 000); co-morbidity with a bleeding disorder; comorbidity with thyroid dysfunction; pregnancy; haemoglobin levels <10 g/dl and haematocrit <30; anaemia on active pharmacological treatment or receiving blood transfusion or steroids;
3. having metastatic or recurrent disease, history of preexisting peripheral neuropa- thy prior to chemotherapy, uncontrolled seizure disorder, unstable cardiac disease or myocardial infarction within 6 months prior to study entry;
4. Being pregnant or nursing, or having used acupuncture for peripheral neuropathy within 6 months prior to study entry;
5. Life expectancy <6 months;
6. Lymphedema of limbs;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
FACT/GOG-Ntx | 6
  Patients self-reported FACT/ GOG-NTX at 6 weeks (end of treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qinghai University, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: No